CLINICAL TRIAL: NCT06873685
Title: Soft Tissue Sarcoma: Instrumented Evaluation of Motor Performance and Impact of Robotic Rehabilitation, Nutrition and Quality of Life Assessment (START-RUN1)
Brief Title: Soft Tissue Sarcoma: Motor Performance, Robotic Rehabilitation, Nutrition, and Quality of Life
Acronym: START-RUN1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FPUCBM_STARTRUN1; PNRR-TR1-2023-12378226 (Other Grant/Funding Number: Ministry of Health, EU-funded, Next Generation EU-PNRR M6C2 - Inv.2.1)
Record Dates: First submitted 2025-02-10; First posted 2025-03-13 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Sarcoma, Soft Tissue
Keywords: rehabilitation; nutrition; quality of life; instrumented assessment of motor performance
MeSH Terms: conditions — Sarcoma | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rehabilitation (Experimental): Conventional and robotic / technological rehabilitation treatments targeting the upper or lower limb, based on tumor location.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — After surgery, patients will undergo a personalized rehabilitation program incorporating both conventional and robotic-based approaches. Depending on tumor location, rehabilitation will focus on either the upper or lower limbs.
  For lower limb rehabilitation, robotic or technological devices will be utilized for gait training with bodyweight support, as well as for balance and proprioception training. Upper limb rehabilitation will involve robotic or sensor-based devices enabling passive, active, and active-assistive movements of the shoulder, elbow, and hand.
  Treatment will be provided in various settings- inpatient, outpatient, or home-based- tailored to each patient's specific needs. Sessions will be conducted daily for 45 minutes, five days per week, over a two-month period.

SUMMARY:
Soft tissue sarcomas are a group of rare and heterogeneous tumors. Surgery is the mainstay of treatment and microscopic negative margins need to be achieved to improve disease local control. We designed this prospective study to evaluate the main features of motor impairment and the impact of tailored robotic rehabilitation techniques in patients treated for localized soft tissue sarcoma (surgery alone, or surgery + radiation or radiochemotherapy). Specific patients' motor strategies will be quantitatively measured through a biomechanical assessment, including the analysis of joint kinematics, and muscle activity timing patterns. Considering the influence of motor impairment after demolitive surgery, a major interest of this study will be focused on nutrition and Quality of life which will be prospectively evaluated by specific questionnaires at different time points.

DETAILED DESCRIPTION:
This is a non-profit, multicenter, non-controlled interventional study aimed at evaluating the main characteristics of motor disability and the impact of personalized robotic rehabilitation in patients undergoing surgical treatment for localized soft tissue sarcoma (STS).

Aim 1: Identify the clinical characteristics and motor deficits following surgical intervention for soft tissue sarcoma (STS).

Aim 2: Evaluate the impact of a personalized robotic rehabilitation treatment on motor recovery in patients with STS.

Aim 3: Assess the impact of perioperative treatments and surgery on quality of life and nutritional status in patients with STS.

The primary endpoint of the study is the assessment of functional deficits and motor quality in patients with STS who have undergone surgical treatment, both after surgery and after a personalized rehabilitation program. The evaluation of functional deficits will include the analysis of functional impairment, activity limitations, and pain, which will be assessed using validated clinical scales. Motor quality will be measured using MIMU and EMG sensors and motor tests to study muscle activity.

The secondary endpoints will include:

1. a comprehensive patient and disease assessment, recording: demographic information and patient characteristics; past medical history; tumor location; histopathological tumor characteristics; details on neoadjuvant therapies and surgical procedures.
2. the Quality of life assessment of the patients;
3. the nutritional status assessment of the patients.

Study Procedures and Interventions:

Comprehensive assessments-including general, clinical, instrumental, quality of life, and nutritional evaluations-will be conducted at:

T0 (at diagnosis) to establish aims to characterize the impact of the tumor on the patient's functional abilities.

T0+ (after radio-chemotherapy, if applicable) to assess the potential effects of radio-chemotherapy before surgery.

Patients eligible for rehabilitation treatment will follow a structured evaluation process:

T1 (within one month after surgery): reassessment to determine the functional impact of surgery.

Rehabilitation phase: Patients will undergo conventional and robotic rehabilitation therapies tailored to the upper or lower limbs.

T2 (after two months of rehabilitation): reassessment to measure functional recovery and rehabilitation outcomes.

T3 (within eight-months from surgery): follow-up.

The sample size was calculated based on a change after the rehabilitation program at least equal to the MCID of the scale. Specifically, 67 individuals are necessary considering a 2-sided, paired t-test, an MCID of 7 points, a common standard deviation of 20 points, a correlation coefficient between paired samples of 0.5, a significance threshold of 0.05, and a power of 0.80. This sample size will be increased to 90 individuals to account for a 25% loss at T2 owing to patients who will be unable to begin the rehabilitation intervention or who will develop clinical complications during the rehabilitation intervention. The power calculation was limited to patients with RPS and lower limb ESTS since the MCID of the TESS for the upper limb module has not been published. Moreover, we will enroll 30 patients with upper limb ESTS, based on number of patients referred and operated at our units (UO1 and UO3) in the last 2 years. Findings achieved in these patients will be considered exploratory for the scanty information currently available in the literature.

All participating centers will follow a standardized operating procedure regarding treatment and outcome assessment to ensure consistency across all sites. Data will be systematically collected using the REDCap (Research Electronic Data Capture) platform.

ELIGIBILITY:
Inclusion Criteria:

1. patient with primary and localized STS who is a candidate for limb-sparing surgery or retroperitoneal multivisceral resection (including partial or complete resection of the iliopsoas muscle with functional loss and potential femoral nerve involvement) with curative intent;
2. age 18 years or older.

Exclusion Criteria:

1. recurrent tumors;
2. metastatic disease;
3. candidate for palliative and non-radical surgery;
4. refusal to sign informed consent;
5. Pregnant or breastfeeding women at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in patients' physical function after the rehabilitation treatment as assessed by the Toronto Extremity Salvage Score (TESS) score | T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment)
  The Toronto Extremity Salvage Scores is the most commonly used, valid, and disease-specific measure to assess physical function in patients with bone and soft tissue tumors of the extremities undergoing limb salvage surgery. The Italian version will be used. The score ranges from 0 to 100, with 100 being the best score. According to tumor's location, either the upper or the lower limb section will be used. We will employ the Italian version of the TESS.

SECONDARY OUTCOMES:
Toronto Extremity Salvage Score (TESS) | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  The Toronto Extremity Salvage Scores is the most commonly used, valid, and disease-specific measure to assess physical function in patients with bone and soft tissue tumors of the extremities undergoing limb salvage surgery. The Italian version will be used. The score ranges from 0 to 100, with 100 being the best score. According to tumor's location, either the upper or the lower limb section will be used. We will employ the Italian version of the TESS.
Musculoskeletal Tumor Society Rating Scale (MSTS) | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  The Musculoskeletal Tumor Society Rating Scale (MSTS) scoring system is a commonly used functional evaluation system for patients who undergo surgery for musculoskeletal tumors. The MSTS system consists of six key criteria, each graded on a five-point scale (0 to 5 points). The total score ranges from 0 to 30 points, where higher scores indicate better functional outcomes. According to tumor's location, either the upper or the lower limb section will be used.
Numerical Pain Rating Scale (NPRS) | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery);T1 (1 months after surgery);T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery).
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale, from 0 (no pain) to 10 (worst pain imaginable).
Brief Pain Questionnaire (BPI) | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery);T1 (1 months after surgery);T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  The Brief Pain Inventory (BPI) is a rapid tool for assessing clinical pain. It consists of two sections. The first section, composed of four items, assesses pain intensity in different situations (current pain, worst pain, least pain, and average pain). The second section examines the impact of pain on daily life through seven items, covering work, recreational activities, mobility, sleep quality, mood, interpersonal relationships, and overall quality of life. Each item is rated using an 11-point Likert scale, ranging from 0 ("no pain/no interference") to 10 ("maximum pain/maximum interference").
Douleur Neuropathique en 4 Questions (DN4) | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery);T1 (1 months after surgery);T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery).
  Douleur Neuropathique en 4 Questions (DN4) questionnaire is a validated clinician-administered screening tool for neuropathic pain. It ranges from 0 to 10; higher values means higher neuropathic pain probability.
Leeds Assessment of Neuropathic Symptoms and Signs Scale (LANSS) | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery);T1 (1 months after surgery);T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery).
  Leeds Assessment of Neuropathic Symptoms and Signs Scale (LANSS) is a simple clinical tool that can be used to identify pain of predominantly neuropathic origin. Contains 5 symptom items and 2 clinical examination items[1]. For the clinical examination, a cotton wool and 23 gauge needle is required. A score of 12 or above is indicative of predominantly neuropathic pain.
Kinematic assessment of motor performance | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery);T1 (1 months after surgery);T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery).
  Patients' motor strategies will be quantitatively measured through a biomechanical assessment using a network of Magneto-Inertial Measurement Unit (MIMU) sensors, to measure joint kinematics, and spatio-temporal parameters.
Surface electromyography (sEMG) assessment | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery);T1 (1 months after surgery);T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery).
  Patients' motor strategies will be quantitatively evaluated using a surface electromyography (sEMG) system, allowing for the analysis of muscle activation timing patterns.
Quality-of-Life Questionnaire (QLQ)-C30 | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery);T1 (1 months after surgery);T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery).
  The European Organization for Research and Treatment of Cancer (EORTC) questionnaire QLQ-C30 version, is a 30-item instrument designed to measure quality of life in all cancer patients. The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Short Form Health Survey 36 (SF-36) - Physical Composite Score (PCS) | T0 (1 week before surgery), T0+ (after after radiochemotherapy, if administered before surgery), T1 (1 months after surgery) and T2 (after 2 months of rehabilitation treatment), T3 (follow up, within 8 months after surgery)
  The Short Form Health Survey 36 (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures. The Physical Component Score (PCS) score is a composite measure that reflects an individual's overall physical health status. It ranges from 0 to 100. Higher scores indicate better physical health and fewer limitations, while lower scores reflect greater physical impairment.
Short Form Health Survey 36 (SF-36) - Mental Composite Score (MCS) | T0 (1 week before surgery), T0+ (after after radiochemotherapy, if administered before surgery), T1 (1 months after surgery) and T2 (after 2 months of rehabilitation treatment), T3 (follow up, within 8 months after surgery)
  The Short Form Health Survey 36 (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures. The Mental Composite Score (MCS) is a composite measure that reflects an individual's overall mental status. It ranges from 0 to 100, with 0 representing the worst possible mental health and 100 representing the best possible mental health..
PREDIMED questionnaire | T0 (1 week before surgery)
  The PREDIMED 14-item questionnaire is a rapid screening tool designed to assess adherence to the Mediterranean diet. Each of the 14 items is a yes/no question, with responses scored as follows: 1 point for a response indicating adherence to a Mediterranean diet principle; 0 points for a response indicating non-adherence. The total score ranges from 0 to 14, with higher scores indicating greater adherence to the Mediterranean diet.
Food diary compilation | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  Patients' compilation of a Food Diary registering 3 non-consecutive days per week ( as for NIH, National Cancer Institute, Dietary assessment Primer)
Weight in kilograms | T0 (1 week before surgery), T0+ (after after radiochemotherapy, if administered before surgery), T1 (1 months after surgery) and T2 (after 2 months of rehabilitation treatment), T3 (follow up, within 8 months after surgery)
  It is a measure of body mass weight expressed in Kg
Height in meters | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  It is a measure of body height expressed in meters.
Body mass Index in kg/(m^2) | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  It is a measure which combines the height and weight values to report Body Mass Index (BMI) expressed in kg/m²; this parameter is valid for adult men and women.
Arm circumferences expressed in cm | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  Measures of arm circumferences expressed in cm.
Waist circumferences expressed in cm | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  Measures of waist circumferences expressed in cm.
Hips circumferences expressed in cm | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  Measures of hips circumferences expressed in cm.
Bioimpedance analysis (BIA) measurements | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  it is a non-invasive measurement of body fat, lean muscle mass and hydration
Concentration of blood levels of haemoglobin in g/dL | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  Blood measurements of haemoglobin (g/dL) measured with colorimetric method.
Concentration of blood levels of lymphocite expressed in count of cells or percentage | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  Blood measurements of total lymphocyte in count of cells or percentage
Concentration of albumine serum levels in g/dL | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  Serum measurements of albumin in g/dL measured with colorimetric method.
Concentration of total cholesterol serum levels in mg/dL | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  Serum measurements of total cholesterol in mg/dL measured with colorimetric method.
Concentration of serum C-reactive protein (CRP) | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  Serum measurements of C-reactive protein mg/dL measured with colorimetric method.
Concentration of glucose serum levels in mg/dL | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  Serum measurements of glucose in mg/dL measured with colorimetric method.
Controlling Nutritional Status (CONUT) | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  The Controlling Nutritional Status (CONUT) is a nutritional scoring tool that is calculated using serum concentration of: albumin, total cholesterol level, total lymphocyte count
Nutritional Risk Index score (NRI) | T0 (1 week before surgery); T0+ (after after radiochemotherapy, if administered before surgery); T1 (1 months after surgery); T2 (after 2 months of rehabilitation treatment); T3 (follow up, within 8 months after surgery)
  The Nutritional Risk Index score (NRI) is a nutritional index calculated from measurements of weight and concentration of serum albumin.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Vincenzi, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario Campus Bio-Medico
Locations (3):
- Italy (3):
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Lazio
  - Fondazione Don Carlo Gnocchi ONLUS, Roma, RM
  - Istituto Nazionale Tumori-IRCCS-Fondazione G.Pascale, Napoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanaka A, Okamoto M, Kito M, Yoshimura Y, Aoki K, Suzuki S, Takazawa A, Komatsu Y, Ideta H, Ishida T, Takahashi J. Muscle strength and functional recovery for soft-tissue sarcoma of the thigh: a prospective study. Int J Clin Oncol. 2023 Jul;28(7):922-927. doi: 10.1007/s10147-023-02348-4. Epub 2023 May 3. PMID 37133781
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] van Eck I, den Hollander D, Desar IME, Soomers VLMN, van de Sande MAJ, de Haan JJ, Verhoef C, Vriens IJH, Bonenkamp JJ, van der Graaf WTA, van Houdt WJ, Husson O. Unraveling the Heterogeneity of Sarcoma Survivors' Health-Related Quality of Life Regarding Primary Sarcoma Location: Results from the SURVSARC Study. Cancers (Basel). 2020 Oct 22;12(11):3083. doi: 10.3390/cancers12113083. PMID 33105807
- [Background] Slump J, Bastiaannet E, Halka A, Hoekstra HJ, Ferguson PC, Wunder JS, Hofer SOP, O'Neill AC. Risk factors for postoperative wound complications after extremity soft tissue sarcoma resection: A systematic review and meta-analyses. J Plast Reconstr Aesthet Surg. 2019 Sep;72(9):1449-1464. doi: 10.1016/j.bjps.2019.05.041. Epub 2019 May 23. PMID 31302071
- [Background] Rossi L, Boffano M, Comandone A, Ferro A, Grignani G, Linari A, Pellegrino P, Piana R, Ratto N, Davis AM. Validation process of Toronto Exremity Salvage Score in Italian: A quality of life measure for patients with extremity bone and soft tissue tumors. J Surg Oncol. 2020 Mar;121(4):630-637. doi: 10.1002/jso.25849. Epub 2020 Jan 19. PMID 31957034
- [Background] Poquet N, Lin C. The Brief Pain Inventory (BPI). J Physiother. 2016 Jan;62(1):52. doi: 10.1016/j.jphys.2015.07.001. Epub 2015 Aug 21. No abstract available. PMID 26303366
- [Background] Pavlidis ET, Pavlidis TE. New trends in the surgical management of soft tissue sarcoma: The role of preoperative biopsy. World J Clin Oncol. 2023 Feb 24;14(2):89-98. doi: 10.5306/wjco.v14.i2.89. PMID 36908679
- [Background] Ogura K, Uehara K, Akiyama T, Shinoda Y, Iwata S, Tsukushi S, Kobayashi E, Hirose T, Yonemoto T, Endo M, Tanzawa Y, Nakatani F, Kawano H, Tanaka S, Kawai A. Minimal clinically important differences in Toronto Extremity Salvage Score for patients with lower extremity sarcoma. J Orthop Sci. 2020 Mar;25(2):315-318. doi: 10.1016/j.jos.2019.03.022. Epub 2019 Apr 16. PMID 31000377
- [Background] McKenzie C, Barker K. Occupational therapy rehabilitation for sarcoma patients following limb salvage surgery: a scoping review. Disabil Rehabil. 2021 Jan;43(2):284-296. doi: 10.1080/09638288.2019.1620874. Epub 2019 Jun 10. PMID 31180732
- [Background] Martinez-Gonzalez MA, Garcia-Arellano A, Toledo E, Salas-Salvado J, Buil-Cosiales P, Corella D, Covas MI, Schroder H, Aros F, Gomez-Gracia E, Fiol M, Ruiz-Gutierrez V, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Munoz MA, Warnberg J, Ros E, Estruch R; PREDIMED Study Investigators. A 14-item Mediterranean diet assessment tool and obesity indexes among high-risk subjects: the PREDIMED trial. PLoS One. 2012;7(8):e43134. doi: 10.1371/journal.pone.0043134. Epub 2012 Aug 14. PMID 22905215
- [Background] Heidari S, Babor TF, De Castro P, Tort S, Curno M. Sex and Gender Equity in Research: rationale for the SAGER guidelines and recommended use. Res Integr Peer Rev. 2016 May 3;1:2. doi: 10.1186/s41073-016-0007-6. eCollection 2016. PMID 29451543
- [Background] Fayers P, Bottomley A; EORTC Quality of Life Group; Quality of Life Unit. Quality of life research within the EORTC-the EORTC QLQ-C30. European Organisation for Research and Treatment of Cancer. Eur J Cancer. 2002 Mar;38 Suppl 4:S125-33. doi: 10.1016/s0959-8049(01)00448-8. PMID 11858978
- [Background] Enneking WF, Dunham W, Gebhardt MC, Malawar M, Pritchard DJ. A system for the functional evaluation of reconstructive procedures after surgical treatment of tumors of the musculoskeletal system. Clin Orthop Relat Res. 1993 Jan;(286):241-6. PMID 8425352
- [Background] Davis AM, Wright JG, Williams JI, Bombardier C, Griffin A, Bell RS. Development of a measure of physical function for patients with bone and soft tissue sarcoma. Qual Life Res. 1996 Oct;5(5):508-16. doi: 10.1007/BF00540024. PMID 8973131
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] Cocks K, Wells JR, Johnson C, Schmidt H, Koller M, Oerlemans S, Velikova G, Pinto M, Tomaszewski KA, Aaronson NK, Exall E, Finbow C, Fitzsimmons D, Grant L, Groenvold M, Tolley C, Wheelwright S, Bottomley A; European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Group. Content validity of the EORTC quality of life questionnaire QLQ-C30 for use in cancer. Eur J Cancer. 2023 Jan;178:128-138. doi: 10.1016/j.ejca.2022.10.026. Epub 2022 Nov 1. PMID 36436330
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Caraceni A, Mendoza TR, Mencaglia E, Baratella C, Edwards K, Forjaz MJ, Martini C, Serlin RC, de Conno F, Cleeland CS. A validation study of an Italian version of the Brief Pain Inventory (Breve Questionario per la Valutazione del Dolore). Pain. 1996 Apr;65(1):87-92. doi: 10.1016/0304-3959(95)00156-5. PMID 8826494
- [Background] Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, Cunin G, Fermanian J, Ginies P, Grun-Overdyking A, Jafari-Schluep H, Lanteri-Minet M, Laurent B, Mick G, Serrie A, Valade D, Vicaut E. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005 Mar;114(1-2):29-36. doi: 10.1016/j.pain.2004.12.010. Epub 2005 Jan 26. PMID 15733628
- [Background] Bennett M. The LANSS Pain Scale: the Leeds assessment of neuropathic symptoms and signs. Pain. 2001 May;92(1-2):147-57. doi: 10.1016/s0304-3959(00)00482-6. PMID 11323136
- [Background] Barnes ME, Elliott JA, McIntyre TV, Boyle EA, Gillis AE, Ridgway PF. Sarcopenia and obesity among patients with soft tissue sarcoma - Association with clinicopathologic characteristics, complications and oncologic outcome: A systematic review and meta-analysis. Eur J Surg Oncol. 2021 Sep;47(9):2237-2247. doi: 10.1016/j.ejso.2021.04.024. Epub 2021 May 20. PMID 34023166
- [Background] Apolone G, Mosconi P. The Italian SF-36 Health Survey: translation, validation and norming. J Clin Epidemiol. 1998 Nov;51(11):1025-36. doi: 10.1016/s0895-4356(98)00094-8. PMID 9817120